CLINICAL TRIAL: NCT05144412
Title: Real-world In-hospital Outcomes and Potential Predictors of Heart Failure in Pregnant Women With Heart Disease in Southwestern China
Brief Title: Pregnant Women With Heart Disease in Southwestern China
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Wei Huang, Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2019XMSB0001234
Record Dates: First submitted 2021-12-01; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Complications of Heart Disease (HD)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Little is known about the status of maternal, obstetric and neonatal complications and the potential predictors of developing heart failure (HF) in the mothers with underlying heart disease (HD) in Southwestern China. Eligible samples were screened from December, 2010 to December, 2019. Maternal clinical characteristics and in-hospital outcomes were collected and compared in women with and without HD, and in HD subtypes: valvular heart disease (VHD), cardiomyopathy, adult congenital heart disease (ACHD), pulmonary hypertension (PH) and other cardiac condition.

DETAILED DESCRIPTION:
Data Source and Study Population We enrolled patients from seven main medical centers in Southwestern China,that was used to characterize outcomes from December 1, 2010 to December 31, 2019. All pregnant women (excluding abortion, nonfirst delivery, multiple births) were eligible for inclusion in the present analysis. Cardiac disease of pregnant woman in the analysis mainly included valvular heart disease (VHD), cardiomyopathy, adult congenital heart disease (ACHD), pulmonary hypertension (PH) and other cardiac conditions (primary arrythmia, coronary heart disease, anemic heart disease, hyperthyroid heart disease and others). Only singleton records with a unique medical identified number were used in our analysis. Patients aged <18 years and those with missing information including unique patient identifiers were excluded. Records with the same date of birth, admission date, discharge date, and facility name were considered as pure duplications, and only one of such records was kept. The data set was analyzed retrospectively, and the informed consent requirement was waived.

Outcome Measures Hypertensive disorders of pregnancy were defined and classified mainly as the following two types from ISSHP (International Society for the Study of Hypertension in Pregnancy) Classification, Diagnosis, and Management Recommendations for International Practice: Hypertension known before pregnancy or present in the first 20 weeks; Hypertension arising de novo at or after 20 weeks.[10] Maternal major adverse cardiac events (MACE) were defined as a composite of arrhythmia, shock, cerebrovascular events, heart failure, respiratory failure, in-hospital death, pulmonary embolism, dissection of any artery.[3, 11, 12] Cardiac procedural intervention was also recorded for patients with and without HD. Non-MACE maternal outcomes included acute renal failure, total hospital charges and hypertensive disorders of pregnancy (all types). Obstetric complications mainly included adherent placenta, abruptio placenta, breech delivery, DIC (disseminated intravascular coagulation), early or threatened labor, known or suspected fetal abnormality, laceration, long labor, placental insufficiency, placenta previa, precipitate labor, premature rupture of membranes, polyhydramnios, postpartum hemorrhage and infection. Neonatal adverse clinical events (NACE) were a composite of fetal death (in utero), neonate death (within 30 days of birth), prematurity (<37 weeks), intrauterine growth restriction, respiratory distress syndrome and intracranial cerebral events. NON-MACE variables including infant of low-birth weight (weight<2500g) and fetal macrosomia (weight>4000g) were also measured. HF was defined in these patients with various underlying heart diseases as a clinical syndrome that was characterized by specific symptoms (dyspnea and fatigue) and signs (of fluid retention, such as edema, rales) as judged by the treating cardiologist according to ACC/AHA guidelines.[13] Information for the present analysis was obtained through review of the institutional database, into which data had been entered on discharge of each patient.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women (excluding abortion, nonfirst delivery, multiple births) were eligible for inclusion in the present analysis. Cardiac disease of pregnant woman in the analysis mainly included valvular heart disease (VHD), cardiomyopathy, adult congenital heart disease (ACHD), pulmonary hypertension (PH) and other cardiac conditions (primary arrythmia, coronary heart disease, anemic heart disease, hyperthyroid heart disease and others). Only singleton records with a unique medical identified number were used in our analysis. Records with the same date of birth, admission date, discharge date, and facility name were considered as pure duplications, and only one of such records was kept.

Exclusion Criteria:

* abortion, nonfirst delivery, multiple births Patients aged <18 years and those with missing information including unique patient identifiers were excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: . All primigravid women (excluding abortion, multiparous women, and multiple births) were eligible for inclusion in the present analysis. The cardiac diseases of a pregnant woman in the analysis included VHD, cardiomyopathy, ACHD, PH, and other cardiac conditions (primary arrythmia, coronary HD, anemic HD, and hyperthyroid HD)
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
maternal, obstetric, and neonatal complications | 2010-2019
  major adverse cardiac events (MACEs), obstetric complications and neonatal adverse clinical events (NACEs)

IPD SHARING:
Plan to Share IPD: Undecided